CLINICAL TRIAL: NCT02264925
Title: Thalamic LFPs and VIM DBS in Essential Tremor: Correlation, Evolution, and Therapeutic Perspectives
Acronym: VIM-CLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: APTES 100 rue boileau 69006 Lyon (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2013/15
Record Dates: First submitted 2014-06-20; First posted 2014-10-15 (Estimated); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Essential Tremor
Keywords: Essential tremor; Deep brain stimulation (DBS); Ventral intermediate Thalamus (VIM); Local field potentials (LFPs); Closed loop therapy
MeSH Terms: conditions — Essential Tremor | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deep Brain Stimulation (Experimental): All of included patients will receive a standard deep brain stimulation of the thalamus in order to reduce their essential tremor
  Interventions: Device: Deep Brain Stimulation with Medtronic Activa PC+S systems

INTERVENTIONS:
Device: Deep Brain Stimulation with Medtronic Activa PC+S systems — Deep Brain Stimulation of VIM.

SUMMARY:
The objective of this study is to characterize through spectral analysis intra-thalamic local field potentials (LFPs) recorded through implanted DBS leads during periods with and without tremor in patients suffering from severe essential tremor.

DETAILED DESCRIPTION:
Essential tremor (ET) is one of the most common adult movement disorders with a prevalence of 4% in the general population. Although several medications (primidone, beta-adrenergic blockers, benzodiazepines…) are commonly used, few of them are truly effective for controlling the severe forms of ET. Since 1987, an alternative has emerged with the development of high frequency deep brain stimulation (DBS) of the thalamic nucleus ventralis intermedius (VIM). This surgical technique now represents the gold standard treatment for tremor-disabled ET patients. Although VIM-DBS is clearly effective for treatment of essential tremor (ET) a partial loss of DBS effectiveness may occur over time in some patients. This loss of DBS effectiveness could be related to an adaptation of the local neuronal network to chronic stimulation (changes in synaptic plasticity). In order to avoid this problem, investigators plan to develop a intermittent mode of VIM stimulation using a new Medtronic device combining a DBS system with local field potential (LFPs) sensing capability. First, investigators propose to analyse VIM LFPs in order to define a tremor biomarker in 10 patients operated for severe ET. Thereafter, investigators will automatically detect this biomarker using a specific algorithm and use it to trigger stimulation at the onset of tremor only. Thus, this project will allow us to optimize DBS therapy in ET, by improving the longevity of implantable devices and avoiding the loss of efficacy previously reported

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from severe and disabling ET with serious impact on their quality of life (QoL).
* 18-70 years old
* Free of evolutive and untreated psychiatric disorder
* Tremor must be predominant in the upper limbs although it can affect the lower limbs, head and voice.
* Affiliation to a social security system
* Written informed consent signed by the participant and the investigator (prior to any examination required by research)

Exclusion Criteria:

* Parkinsonian tremor
* Pregnancy or lactating women
* Severe co-morbidity (cardiac, renal or respiratory failures, evolutive cancer)
* Impaired cognitive functions (score <130 on Mattis scale).
* Patients with severe atrophy or lesions on MRI
* Depression (Beck > 10)
* Participation in another clinical research for 18 months (after surgery)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
LFPs records 3 month after implantation | 3 month after implantation
  in order to characterize the features of tremor-related thalamic activity during the initiation of movement-related tremor-induced activity
LFPs records 12 month after implantation | 12 month after implantation
  in order to characterize the features of tremor-related thalamic activity during the initiation of movement-related tremor-induced activity

CONTACTS AND LOCATIONS:
Overall Officials: BURBAUD Pierre, MD-PhD, Study Director — University Hospital Bordeaux, France; Nicolas LANGBOUR, PhD, Study Chair — IMN CNRS UMR 5293, Université Bordeaux 2 Segalen
Locations (1):
- University Hospital Bordeaux, France, Bordeaux, France

REFERENCES:
- [Background] Barbe MT, Liebhart L, Runge M, Pauls KA, Wojtecki L, Schnitzler A, Allert N, Fink GR, Sturm V, Maarouf M, Timmermann L. Deep brain stimulation in the nucleus ventralis intermedius in patients with essential tremor: habituation of tremor suppression. J Neurol. 2011 Mar;258(3):434-9. doi: 10.1007/s00415-010-5773-3. Epub 2010 Oct 8. PMID 20927533
- [Background] Benabid AL, Pollak P, Louveau A, Henry S, de Rougemont J. Combined (thalamotomy and stimulation) stereotactic surgery of the VIM thalamic nucleus for bilateral Parkinson disease. Appl Neurophysiol. 1987;50(1-6):344-6. doi: 10.1159/000100803. PMID 3329873
- [Background] Blomstedt P, Hariz GM, Hariz MI, Koskinen LO. Thalamic deep brain stimulation in the treatment of essential tremor: a long-term follow-up. Br J Neurosurg. 2007 Oct;21(5):504-9. doi: 10.1080/02688690701552278. PMID 17922323
- [Background] Brown P, Williams D. Basal ganglia local field potential activity: character and functional significance in the human. Clin Neurophysiol. 2005 Nov;116(11):2510-9. doi: 10.1016/j.clinph.2005.05.009. Epub 2005 Jul 18. PMID 16029963
- [Background] Garcia Ruiz P, Muniz de Igneson J, Lopez Ferro O, Martin C, Magarinos Ascone C. Deep brain stimulation holidays in essential tremor. J Neurol. 2001 Aug;248(8):725-6. doi: 10.1007/s004150170127. No abstract available. PMID 11569910
- [Background] Hariz MI, Shamsgovara P, Johansson F, Hariz G, Fodstad H. Tolerance and tremor rebound following long-term chronic thalamic stimulation for Parkinsonian and essential tremor. Stereotact Funct Neurosurg. 1999;72(2-4):208-18. doi: 10.1159/000029728. PMID 10853080
- [Background] Limousin P, Speelman JD, Gielen F, Janssens M. Multicentre European study of thalamic stimulation in parkinsonian and essential tremor. J Neurol Neurosurg Psychiatry. 1999 Mar;66(3):289-96. doi: 10.1136/jnnp.66.3.289. PMID 10084526
- [Background] Schuurman PR, Bosch DA, Bossuyt PM, Bonsel GJ, van Someren EJ, de Bie RM, Merkus MP, Speelman JD. A comparison of continuous thalamic stimulation and thalamotomy for suppression of severe tremor. N Engl J Med. 2000 Feb 17;342(7):461-8. doi: 10.1056/NEJM200002173420703. PMID 10675426
- [Background] Stacy MA, Elble RJ, Ondo WG, Wu SC, Hulihan J; TRS study group. Assessment of interrater and intrarater reliability of the Fahn-Tolosa-Marin Tremor Rating Scale in essential tremor. Mov Disord. 2007 Apr 30;22(6):833-8. doi: 10.1002/mds.21412. PMID 17343274
- [Background] Yoshida F, Martinez-Torres I, Pogosyan A, Holl E, Petersen E, Chen CC, Foltynie T, Limousin P, Zrinzo LU, Hariz MI, Brown P. Value of subthalamic nucleus local field potentials recordings in predicting stimulation parameters for deep brain stimulation in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2010 Aug;81(8):885-9. doi: 10.1136/jnnp.2009.190918. Epub 2010 May 12. PMID 20466699